CLINICAL TRIAL: NCT02723357
Title: The Impact of Family Financial Support on Parental Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Adam Schickedanz, Clinical Instructor and Clinical Scholar, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UCLASchickedanzFCMH
Record Dates: First submitted 2016-03-24; First posted 2016-03-30 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Financial Coaching; Mental Disorders; Social Determinants; Medical-Financial Partnership; Toxic Stress
Keywords: Financial Coaching; Mental Health; Social Determinants; Medical-Financial Partnership; Toxic Stress
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Financial Coaching & Access to Services (Experimental): Participants in this arm will receive monthly financial coaching and access to basic social service referrals until either one year, closure of all financial needs, or loss to follow up.
  Interventions: Behavioral: Financial Coaching; Behavioral: Access to Social Service Referrals
- Access to Services (Active Comparator): Participants in this arm will receive access to basic social service referrals until either one year, closure of all financial needs, or loss to follow up.
  Interventions: Behavioral: Access to Social Service Referrals

INTERVENTIONS:
Behavioral: Financial Coaching — Enrollment in one-to-one financial coaching intervention to support savings, income, and credit while reducing debt using available tools in the community development field.
  Arms: Financial Coaching & Access to Services
Behavioral: Access to Social Service Referrals — Access to referrals for common social needs.

SUMMARY:
The investigators have partnered with financial coaching organizations to establish what the investigators have termed a "Medical-Financial Partnership (MFP)" that offers financial coaching to improve financial and mental health. The investigators will evaluate the MFP's impact on mental health using the Kessler-6 emotional distress scale.

DETAILED DESCRIPTION:
Financial coaching is a new tool in the field of community development, but it has already demonstrated significant financial impact in a number of studies, including one randomized trial conducted by the Urban Institute. Financial coaching improves participant financial literacy, budgeting, saving for financial emergencies, and debt level. The investigators' project will help clinicians and the field of community economic development understand health and well-being through a new economic lens and assess the health-related impacts of the emerging field of financial coaching. The investigators have partnered with financial coaching organizations to establish what they have termed a "Medical-Financial Partnership (MFP)" that offers financial coaching to improve financial and mental health. The investigators will evaluate the MFP's impact on mental health using the Kessler-6 emotional distress scale as the outcome variable.

Community-based participants will be recruited from South Los Angeles and randomized to receive either monthly financial coaching plus access to referral for social services (intervention) or access to referral for social services alone (control). Inclusion criteria include having dependents under age 18, having some form of income, and having a tax identification number (social security number or Individual Tax Identification Number). Participants will be surveyed quarterly regarding their mental health using the Kessler-6 emotional distress scale.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers/Parents with one or more child dependents, income of any sort, and a tax identification number.

Exclusion Criteria:

* Inability to partake in financial coaching due to physical limitations or primary language other than Spanish or English.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Mental Health | Up to one year (if possible)
  Mental health as assessed by the Kessler-6 scale of emotional distress

CONTACTS AND LOCATIONS:
Overall Officials: Adam Schickedanz, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- LIFT-LA in Affiliation with UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No